CLINICAL TRIAL: NCT00759109
Title: Long-term Pegylated Alfa-2b Interferon Therapy of Patients With Hepatitis C-related Cirrhosis and High Liver Cell Proliferation: a Multicenter Study of Hepatocellular Carcinoma Prevention in Patients Non-responders to Combined Therapy With Alpha Interferon + Ribavirin or Peginterferon Alpha + Ribavirin or to Interferon Monotherapy
Brief Title: Pegylated Alfa-2b Interferon Therapy of Patients With Hepatitis C-related Cirrhosis and High Liver Cell Proliferation (P02733/MK-4031-085)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P02733
Record Dates: First submitted 2008-08-26; First posted 2008-09-25 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — peginterferon alfa-2b; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A - PegIntron (Experimental): Participants randomized to Arm A received peginterferon α-2b (PegIntron), 50 μg, weekly, subcutaneously (SC), for a period of 3 years.
  Interventions: Biological: Peginterferon alfa-2b
- Arm B - Control (Other): Participants randomized to Arm B were under observation and received no treatment.
  Interventions: Other: Observation (no treatment)

INTERVENTIONS:
Biological: Peginterferon alfa-2b — Peginterferon alfa-2b, 50 μg, weekly, SC, for a period of 3 years.
  Other Names: PegIntron; Pegylated Alfa-2b; SCH 054031
  Arms: Arm A - PegIntron
Other: Observation (no treatment) — No treatment was given to participants enrolled in the control arm (Arm B).
  Arms: Arm B - Control

SUMMARY:
This study aims to compare the role of peginterferon α-2b (50 μg/week) vs. control (no treatment) in the prevention of hepatocellular carcinoma, in adult patients with cirrhosis and initial signs of portal hypertension who did not respond to previous combined therapy with interferon alfa + ribavirin or peginterferon alfa + ribavirin or to interferon alfa monotherapy and with a high proliferation rate before entering the study. The duration of treatment will be 3 years, and the follow-up period will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic participants, both sexes, Child Pugh A, B, HCV-RNA positive, age < 70 years
* Participants non-responders to IFN + Ribavirin or PegIFN + Ribavirin or IFN monotherapy
* Pre-therapy liver biopsy (< 36 months) with PCNA-LI > 2.0
* Fibrosis score 5-6 (Ishak)
* Initial portal hypertension, such as gastroesophageal varices or one of the following US sign:

  * Collateral circles
  * Spleen longitudinal diameter > 12 cm
  * Portal vein diameter at hilus > 12 mm
  * Portal flow > 12 cm/sec
  * Participants must have the following minimum hematologic and biochemical criteria:
  * Hemoglobin >= 11 g/dL
  * Granulocyte count > 1,000/mm^3
  * Platelets > 70,000/mm^3
  * Prothrombin activity > 50%
  * Total bilirubin <3 mg/dL
  * Albumin >= 3.5 g/dL
  * Serum creatinine within normal limits
* Uric Acid within normal limits
* Thyroid Stimulating Hormone (TSH), within normal limits
* Antinuclear antibodies (ANA) < 1:160
* Written informed consent
* Women of childbearing potential must have a negative pregnancy test
* Acceptance of patients of both sexes of proper contraceptive measures for the study period

Exclusion Criteria:

* Pregnant or breast-feeding women
* Co-infection with HIV and/or HBV
* Autoimmune hepatitis or history of autoimmune disease
* Alcoholic liver disease
* Metabolic disease
* HCC
* Participants with liver and kidney transplants
* Evidence of decompensated liver disease such as history or presence of ascites, bleeding varices, spontaneous encephalopathy
* Chronic renal failure or creatinine clearance < 50 mL/min
* Pre-existing thyroid disease unless it can be controlled with conventional treatment
* History or presence of psychiatric condition, especially depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt
* Epilepsy and/or compromised central nervous system (CNS) function
* Significant cardiovascular dysfunction within the previous 6 months before the study starts (eg, angina, congestive heart failure, recent myocardial infarction, moderate or severe hypertension, significant arrhythmia)
* Hemoglobinopathies
* Poorly controlled diabetes mellitus
* Chronic pulmonary disease (eg, chronic obstructive pulmonary disease)
* Clinical gout
* Hypersensitivity to interferons or any component of the drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Intent-to-Treat (ITT) population included all randomized participants who took at least one dose of medication, and presented at least one further efficacy evaluation. No efficacy assessment post-baseline was obtained for 4 participants in the control group, therefore the ITT population included 146 (74 PegIntron + 72 Control) participants.
Groups:
- Arm A - PegIntron: Participants randomized to Arm A received peginterferon α-2b, 50 μg, weekly, for a period of 3 years.
Period: Overall Study
Arm/Group | Arm A - PegIntron | Arm B - Control
Started | 74 | 76
Completed | 35 (From both arms combined, 7 discontinued due to death and there were 8 deaths during follow up.) | 41 (From both arms combined, 7 discontinued due to death and there were 8 deaths during follow up.)
Not Completed | 39 | 35
Not completed — Adverse Event | 17 | 12
Not completed — Inability to comply | 1 | 1
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 4 | 6
Not completed — Started new therapy | 2 | 6
Not completed — HCV RNA negative | 1 | 0
Not completed — Participant moved to a different city | 0 | 1
Not completed — Participant had a liver transplant | 0 | 1
Not completed — Lost during study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - PegIntron | Arm B - Control | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] — ITT Population
  Years | 57 (8.7) | 59.7 (7.2) | 58.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT Population
  Participants
    Female | 22 | 34 | 56
    Male | 52 | 38 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Development of Hepatocellular Carcinoma (HCC)
Description: Participants were tested for focal lesions by liver ultrasound and for AFP levels every 6 months the during study (treatment and follow-up).
  The development of hepatocellular carcinoma was determined by:
  1. the appearance of a focal lesion detected by liver ultrasound with metastases confirmed by fine needle biopsy, or
  2. the appearance of a focal lesion detected by ultrasound + alphafetoprotein (AFP) levels in blood >400 ng/mL.
Time Frame: During 3 years of treatment and 2 years of follow-up
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Arm A - PegIntron | Arm B - Control
Number analyzed (Participants) | 74 | 72
Participants | 15 | 11

2. Secondary Outcome: Number of Participants With Development of Hepatic Decompensation
Description: The development of hepatic decompensation, defined as worsening of the hepatic function as measured by Child Pugh Score. The Child Pugh score was calculated based on biochemical changes (changes in serum albumin, serum bilirubin, prothrombin time) and clinical impairment (ascites, encephalopathies) or both. Each of the 5 parameters was scored from 1-3, and the Child Pugh Score represented the total score. The maximum score was 15, and a score of 10-15 represents the worst outcome and a life expectancy of 1-3 years.
Time Frame: Baseline, During 3 years of treatment and 2 years of follow-up
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Arm A - PegIntron | Arm B - Control
Number analyzed (Participants) | 74 | 72
Participants | 4 | 9

3. Secondary Outcome: Survival Time of Participants
Description: Survival time was defined as time from screening visit to the death of the participant and was studied with Kaplan-Meier and Log-rank tests. If a participant did not die, he or she was censored with the last available date.
Time Frame: During 3 years of treatment and 2 years of follow-up
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Arm A - PegIntron | Arm B - Control
Number analyzed (Participants) | 74 | 72
Years | 5.2840 [3.0116 to 5.2841] | 4.0602 [NA to NA] — The median confidence interval for control group could not be calculated due to the low number of events, however, the median survival time for the control group was estimated to be higher than 4.0602 years.

4. Secondary Outcome: Number of Patients With a Virological Response Rate
Description: Virological Response rate was measured by the disappearance of Hepatitis C Virus from serum. Serum samples from participants were analyzed for the
  presence of HCV-RNA using a qualitative polymerase chain reaction (PCR).
Time Frame: Baseline and every year during 3 years of treatment
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Arm A - PegIntron | Arm B - Control
Number analyzed (Participants) | 74 | 72
Participants
  Baseline | 0 | 0
  1 year | 3 | 0
  2 years | 1 | 0
  3 years | 0 | 0

5. Secondary Outcome: Change in the Proliferating Cell Nuclear Antigen Labeling Index (PCNA-LI)
Description: PCNA-LI was measured at baseline and at 18 months of treatment, and the change in PCNA-LI was calculated.
  To measure PCNA-LI, liver tissue samples obtained from biopsies were fixed and immunostained to detect PCNA. PCNA-LI is the percentage of immunohistochemically stained (PCNA positive) cells in 1,000 HCC cells counted. A higher PCNA-LI indicates a worse outcome.
Time Frame: Baseline and at 18 months of treatment
Population: Participants with tissue biopsies at 18 months.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A - PegIntron | Arm B - Control
Number analyzed (Participants) | 37 | 26
Score on a scale | -2.0 (3.2) | -0.9 (2.4)

6. Other Pre Specified Outcome: Proliferating Cell Nuclear Antigen Labeling Index (PCNA-LI) at Baseline
Description: Liver tissues obtained from biopsies were fixed and immunostained to detect PCNA. PCNA-LI is the percentage of immunohistochemically stained (PCNA positive) cells in 1,000 HCC cells counted. A higher PCNA-LI indicates a worse outcome.
Time Frame: Baseline
Population: ITT population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A - PegIntron | Arm B - Control
Number analyzed (Participants) | 74 | 72
Score on a scale | 4.2 (2.1) | 3.9 (1.6)

ADVERSE EVENTS:
Description: A total of 15 serious adverse events resulted in death.
Arm/Group | Arm A - PegIntron | Arm B - Control
Serious Adverse Events (participants affected / at risk) | 36/74 | 30/76
Other Adverse Events (participants affected / at risk) | 55/74 | 36/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - PegIntron (N=74) | Arm B - Control (N=76)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 2 (2) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTRIC DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0)
HYPERPYREXIA (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (2)
BILIARY DILATATION (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2) | 1 (1)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 (1) | 0 (0)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CRYOGLOBULINAEMIA (Immune system disorders) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (2) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
MUSCLE ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS BACTERIAL (Infections and infestations) | 1 (1) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ULTRASOUND LIVER ABNORMAL (Investigations) | 1 (1) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 11 (11)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRAIN MASS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 4 (4) | 0 (0)
COMA HEPATIC (Nervous system disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 2 (2) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0)
QUADRIPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
ANURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
COLON POLYPECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTRECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
BLEEDING VARICOSE VEIN (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
SYSTOLIC HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - PegIntron (N=74) | Arm B - Control (N=76)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 5 (6)
ASCITES (Gastrointestinal disorders) | 1 (1) | 7 (10)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 5 (5)
GASTRITIS (Gastrointestinal disorders) | 3 (4) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 2 (3)
ASTHENIA (General disorders) | 21 (22) | 7 (7)
INFLUENZA LIKE ILLNESS (General disorders) | 20 (23) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 5 (5) | 7 (9)
PYREXIA (General disorders) | 7 (10) | 2 (3)
WEIGHT DECREASED (Investigations) | 6 (6) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
HEADACHE (Nervous system disorders) | 11 (15) | 0 (0)
DEPRESSION (Psychiatric disorders) | 6 (6) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (5)
HYPERTENSION (Vascular disorders) | 5 (6) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the principal investigator (PI) is that the PI agrees not to publish or publicly present any results of the study without the prior written permission of the sponsor. The PI further agrees to allow the sponsor to review, 30 days prior to submission for publication or presentation, copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the study.